CLINICAL TRIAL: NCT04293458
Title: A Multicenter, Single-Arm Study of the Efficacy of EsoGuard(TM) on Samples Collected Using EsoCheck(TM) Versus Esophagogastroduodenoscopy for the Diagnosis of Barrett's Esophagus in an At-Risk Screening Population
Brief Title: Efficacy of EsoGuard on Samples Collected Using EsoCheck Versus EGD for the Diagnosis of BE
Acronym: ESOGUARDBE1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lucid Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Organization: PAVmed Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PR-0139 / EG-CL-101
Record Dates: First submitted 2020-02-26; First posted 2020-03-03 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Barrett Esophagus; Esophageal Adenocarcinoma; Barretts Esophagus With Dysplasia; Barrett's Esophagus Without Dysplasia
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Intervention Model Description: Multicenter, Single Arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- EsoCheck vs. EGD with or without biopsies (Experimental): All subjects will undergo both the EsoCheck (non-invasive esophageal cell sample collection) followed by EGD (with or without biopsies)
  Interventions: Device: EsoGuard

INTERVENTIONS:
Device: EsoGuard — EsoGuard assay (LDT) will be used on cells collected using EsoCheck (510K cleared esophageal cell collection device) and compared to results of EGD plus biopsies (when taken)

SUMMARY:
The study will assess the performance of the combined system, i.e., the use of the EsoGuard assay on cells collected using the EsoCheck 510(k) cleared device, to detect Barrett's Esophagus, with and without dysplasia, and/or Esophageal Adenocarcinoma, in individuals deemed to be at high risk for these conditions (i.e., screening) per ACG guidelines.

DETAILED DESCRIPTION:
This is a multicenter, single-arm study designed to assess the operating characteristics of the EsoGuard diagnostic assay performed on distal esophageal mucosal cells collected using the EsoCheck cell collection device, compared to the gold standard, for the screening of BE with and without dysplasia and for esophageal adenocarcinoma (EAC), in patients at high risk for BE and for whom a screening EGD is indicated according to ACG-established criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged 50 years old and older
2. ≥5 years either of

   * GERD symptoms,
   * GERD treated with proton pump inhibitor (PPI) therapy (whether symptom control is achieved or not), or,
   * any combination of treated and untreated periods, as long the cumulative total is at least 5 years
3. No solid foods eaten for at least 2 hours prior to EsoCheck procedure
4. One or more of the following risk factors:

   1. Caucasian race
   2. Current or past history of cigarette smoking
   3. BMI of at least 30 kg/m2
   4. First-degree relative with BE or EAC

      -

Exclusion Criteria:

1. History of prior EGD procedure
2. Inability to provide written informed consent
3. On anti-coagulant drug(s) that cannot be temporarily discontinued
4. Known history of esophageal varices or esophageal stricture
5. Any contraindication, as deemed in Investigator's medical judgment, to undergoing the EsoCheck procedure, undergoing the EGD procedure, and/or having biopsies taken, including but not limited to due to comorbidities such as coagulopathy or a known history of esophageal diverticula, esophageal fistula and/or esophageal ulceration
6. History of difficulty swallowing (dysphagia) or painful swallowing (odynophagia), including swallowing pills
7. Oropharyngeal tumor
8. History of esophageal or gastric surgery, with exception of uncomplicated surgical fundoplication procedure
9. History of myocardial infarction or cerebrovascular accident within past 6 months
10. History of esophageal motility disorder
11. Currently implanted Linx device

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy | Cross-sectional point in time per subject through study completion which is up to approximately 5 weeks
  The sensitivity and specificity of EsoGuard for the diagnosis of BE on samples collected using EsoCheck, wherein the definitive diagnosis of BE is made by concomitant EGD and biopsy.

SECONDARY OUTCOMES:
Secondary Efficacy | Cross-sectional point in time per subject through study completion which is up to approximately 5 weeks
  Negative predictive value (NPV) and positive predictive value (PPV), calculated for the observed prevalence and over a range of prevalences from 1 to 15%.

OTHER OUTCOMES:
Safety of EsoCheck device administration | Cross-sectional point in time per subject through study completion which is up to approximately 5 weeks
  Assessed by evaluation of AEs/SAEs/ADEs/SADEs/USADEs and Medical Device Deficiency Incidents

CONTACTS AND LOCATIONS:
Overall Officials: Michelle McDermott, Study Director — Lucid Diagnostics
Locations (26):
- United States (23):
  - Lucid Investigative Site, Orange, California
  - Lucid Investigative Site, Englewood, Colorado
  - Lucid Investigative Site, Naples, Florida
  - Lucid Investigative Site, Palm Harbor, Florida
  - Lucid Investigative Site, Macon, Georgia
  - Lucid Investigative Site, Idaho Falls, Idaho
  - Lucid Investigative Site, Rockford, Illinois
  - Lucid Investigative Site, New Orleans, Louisiana
  - Lucid Investigative Site, Shreveport, Louisiana
  - Lucid Investigative Site, Wyoming, Michigan
  - Lucid Investigative Site, Flowood, Mississippi
  - Lucid Investigative Site, Omaha, Nebraska
  - Lucid Investigative Site, New York, New York
  - Lucid Investigative Site, Rochester, New York
  - Lucid Investigative Site, Chapel Hill, North Carolina
  - Lucid Investigative Site, Oklahoma City, Oklahoma
  - Lucid Investigative Site, Philadelphia, Pennsylvania
  - Lucid Investigative Site, Greenville, South Carolina
  - Lucid Investigative Site, Knoxville, Tennessee
  - Lucid Investigative Site, Nashville, Tennessee
  - Lucid Investigative Site, Houston, Texas
  - Lucid Investigative Site, Salt Lake City, Utah
  - Lucid Investigative Site, Richmond, Virginia
- Spain (3):
  - Lucid Investigative Site, Madrid
  - Lucid Investigative Site, Valladolid
  - Lucid Investigative Site, Zaragoza

IPD SHARING:
Plan to Share IPD: No